CLINICAL TRIAL: NCT06287307
Title: Semaglutide 2.4mg for Low Responders After Bariatric Surgery
Acronym: SEABAR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Nederlandse Obestias Kliniek (NOK) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NOK000024
Record Dates: First submitted 2023-06-15; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Obesity, Morbid; Weight Gain
Keywords: Obesity; Semaglutide; GLP-1; Bariatric Surgery; Weight Loss
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Gain; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide 2.4mg (Active Comparator): Patients in this group will receive the active comparator semaglutide 2.4mg. This is a medication which is distributed by an intramuscular injection once weekly.
  Interventions: Drug: Semaglutide 2.4 MG/0.75 ML Subcutaneous Solution [WEGOVY]
- Placebo (Placebo Comparator): Patients in this group will receive the placebo. This is a placebo which is distributed by an intramuscular injection once weekly.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — The placebo will be used in the allocated group in addition to our lifestyle program for the duration of 68 weeks in total.
  Arms: Placebo
Drug: Semaglutide 2.4 MG/0.75 ML Subcutaneous Solution [WEGOVY] — The semaglutide will be used in the allocated group in addition to our lifestyle program for the duration of 68 weeks in total.
  Other Names: Wegovy; Semaglutide
  Arms: Semaglutide 2.4mg

SUMMARY:
In 20 - 30% of the patients, the low responders, sufficient weight loss is not achieved after bariatric surgery. Secondary and/or tertiary bariatric procedures can lead to successful weight loss and resolution of comorbid conditions though, morbidity and mortality rates of these procedures are high. Therefore, additional pharmacotherapy has been suggested. Semaglutide is one of the medications that might improve outcome in the post-bariatric population. Semaglutide is a Glucagon-like peptide-1 (GLP-1) receptor analogue developed to treat type 2 diabetes. It causes glucose-dependent insulin secretion, promotes satiety and inhibits glucagon secretion. In obese (non-bariatric) patients, semaglutide has shown to improve glycemic control, decrease blood pressure, lower cardiovascular risk, and decrease body weight.

DETAILED DESCRIPTION:
The treatment of obesity can be divided into three different fields: non-surgical interventions (e.g. endoscopic techniques, swallowable gastric balloon), pharmacological, and surgical treatment. All these different fields have, as their cornerstone of treatment, lifestyle interventions. Lifestyle interventions have an emphasis on regulation of energy intake and improvement of physical activity. All treatment options are adjunct to the lifestyle interventions. Besides, not all overweight or obese people are eligible for all types of treatment. For instance, pharmacological treatment options are advised in patients with a Body Mass Index (BMI) ≥ 30kg/m2 or a BMI ≥ 27kg/m2 with an obesity-related comorbidity, such as hypertension or diabetes mellitus. Several pharmaceutical agents have been developed for treatment of obesity. These medications generally affect appetite and cause weight loss only when the agent is taken in adjunct to lifestyle modification. Mean weight loss with pharmacological treatment ranges between 4.4 and 14.3%, depending on type of medication and treatment regime.

Bariatric surgery, also called metabolic surgery, includes a variety of surgical procedures in which the gastro-intestinal tract is altered. The most performed types of surgery are the Sleeve Gastrectomy (SG) and the Roux-en-Y gastric bypass (RYGB). All types of surgery cause changes in gut hormones, bile acids and microbiota, which subsequently induce changes in appetite and energy expenditure and thereby causing weight loss. Surgery is generally advised to patients with a BMI ≥ 40kg/m2 or a BMI ≥ 35kg/m2 with comorbid conditions. Compared to lifestyle intervention programs, bariatric surgery has proven to be a superior treatment for morbid obesity. Total weight loss (TWL) is about 20 - 30 %. In addition, bariatric surgery positively influences comorbid conditions, like type 2 diabetes, hypertension, cancer incidence, cardiovascular events and cardiovascular deaths. Thus, currently, bariatric surgery is the most effective treatment for morbid obesity.

However, there is a significant proportion of patients who do not reach "successful" weight loss after bariatric surgery. These patients can be divided in patients who do not reach sufficient weight loss, low responders, and patients who experience weight regain. Although there is no guideline to define who are low responders and what is significant weight regain, unsuccessful weight loss seems to occur in about 20-30% of the population. One of the best predictors of low weight loss in the long-term after surgery is 3-month weight loss. Therefore, this study's clinic provides an extra intervention for the patients who are considered low responders at the 3-month follow-up moment after surgery. The NOK defines a low responder by percentage total weight loss (%TWL) at the 3-month follow-up moment compared to expected weight loss. When %TWL is below the 25% quartile of expected weight loss the patient is considered a low responder. The expected weight loss is determined based on this clinics database of previous patients with the same baseline Body Mass Index (BMI above or below 50 kg/m2), gender and type of surgery. Thus, in the current treatment program patients have a medical consultation in which weight loss is determined three months after surgery. Based on baseline weight and exact number of days after surgery it is calculated whether the patient is a low responder with respect to a private database (currently about 6000 patients). If a patient is considered a low responder then the patient will receive three extra counselling sessions focusing on improving weight loss outcome. This extra intervention is called the plus module and is an addition to the standard program, which consists of multidisciplinary group counselling before and after surgery.

Secondary and/or tertiary bariatric procedures are performed in up to 25% of the patients with unsuccessful weight loss. Although additional surgery can lead to successful weight loss and resolution of comorbid conditions, morbidity and mortality rates of these procedures are higher. Therefore, attention has been focused on pharmacological treatment as an addition to bariatric surgery.

One of the agents that has been suggested for additional pharmacological treatment is semaglutide. Semaglutide is a Glucagon-like peptide-1 (GLP-1) receptor analogue which was initially developed to treat type 2 diabetes. GLP-1 is one of the incretins, a peptide hormone which is normally secreted from L cells in the distal ileum and colon. When secreted, GLP-1 causes an increase in insulin secretion of the beta-cells of the pancreas and a decrease of glucagon production of the alfa-cells. These changes cause a decrease of fasting and post prandial plasma glucose. In addition, GLP-1 also causes delayed gastric emptying. In non-bariatric patients, semaglutide has shown to improve glycaemic control, decrease blood pressure, lower cardiovascular risk and decrease body weight up to one year.

In this trial the effect of semaglutide 2.4 mg once weekly to the plus module for low responders on the improvement of weight loss compared to patient solely receiving the plus module will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* BMI before surgery was ≥ 35.0 kg/m2
* Patient is treated with group consultation at the NOK
* Patient has undergone a primary (banded) RYGB or (banded) sleeve gastrectomy (SG)
* Patient is in the lowest %TWL quartile, 3 months after surgery and will be enrolled in the plus module.

Exclusion Criteria:

* Gastropareses or gastro-intestinal complaints after bariatric surgery
* Type 1 or type 2 diabetes and/or diabetic retinopathy
* Decreased renal function (creatinine clearance < 30 ml/min)
* Liver failure (all)
* Congestive heart failure or angina pectoris NYHA class III and IV
* Malignancy in history
* Pancreatitis (in history)
* (expected) Pregnancy / breast-feeding
* Inflammatory Bowel Disease
* Thyroid malignancy in history
* Use of warfarin or other coumarin derivates

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Weight change from start study at 3 months post operative until 15 months later | 15 months
  To study the weight change from 3 until 18 months after surgery (% total weight loss, TWL) in low responders after bariatric surgery who are treated with Semaglutide 2.4 mg and a lifestyle intervention
Difference between placebo group and treatment group in weight change | 15 months
  compare change in weight to patients receiving placebo and a lifestyle intervention

SECONDARY OUTCOMES:
Weight loss 3 months after surgery | 3 months
  To study the weight loss at 3 months after surgery (before semaglutide start)
Weight loss 6 months after surgery | 6 months
  To study the weight loss at 6 months after surgery (3 months after semaglutide start)
Weight loss 12 months after surgery | 12 months
  To study the weight loss at 12 months after surgery (9 months after semaglutide start)
Weight loss 18 months after surgery | 18 months
  To study the weight loss at18 months after surgery (15 months after semaglutide start)
Metabolic health before surgery (bloodpressure) | Screening for surgery
  To study metabolic health before surgery (before semaglutide start) by using the following parameter: bloodpressure in mmHg
Metabolic health before surgery (HbA1c) | Screening for surgery
  To study metabolic health before surgery (before semaglutide start) by using the following parameter: HbA1c in mmol/mol
Metabolic health before surgery (glucose) | Screening for surgery
  To study metabolic health before surgery (before semaglutide start) by using the following parameter: glucose in mmol/l
Metabolic health before surgery (triglyceride) | Screening for surgery
  To study metabolic health before surgery (before semaglutide start) by using the following parameter: triglycerides in mmol/l
Metabolic health before surgery (LDL) | Screening for surgery
  To study metabolic health before surgery (before semaglutide start) by using the following parameter: LDL in mmol/l
Metabolic health before surgery (HDL) | Screening for surgery
  To study metabolic health before surgery (before semaglutide start) by using the following parameter: HDL in mmol/l
Metabolic health before surgery (total cholesterol) | Screening for surgery
  To study metabolic health before surgery (before semaglutide start) by using the following parameter: total cholesterol in mmol/l
Metabolic health 3 months after surgery (Bloodpressure) | 3 months
  To study metabolic health 3 months after surgery (at semaglutide start) by using the following parameter: bloodpressure in mmHg
Metabolic health 3 months after surgery (HbA1c) | 3 months
  To study metabolic health 3 months after surgery (at semaglutide start) by using the following parameter: HbA1c mmol/mol
Metabolic health 3 months after surgery (glucose) | 3 months
  To study metabolic health 3 months after surgery (at semaglutide start) by using the following parameter: glucose in mmol/l
Metabolic health 3 months after surgery (triglyceride) | 3 months
  To study metabolic health 3 months after surgery (at semaglutide start) by using the following parameter: triglycerides in mmol/l
Metabolic health 3 months after surgery (LDL) | 3 months
  To study metabolic health 3 months after surgery (at semaglutide start) by using the following parameter: LDL in mmol/l
Metabolic health 3 months after surgery (HDL) | 3 months
  To study metabolic health 3 months after surgery (at semaglutide start) by using the following parameter: HDL in mmol/l
Metabolic health 3 months after surgery (total cholesterol) | 3 months
  To study metabolic health 3 months after surgery (at semaglutide start) by using the following parameter: total cholesterol in mmol/l
Metabolic health at 6 months after surgery (bloodpressure) | 6 months
  To study metabolic health 6 months after surgery (3 after semaglutide start) by using the following parameter: bloodpressure in mmHg
Metabolic health at 6 months after surgery (HbA1c) | 6 months
  To study metabolic health 6 months after surgery (3 after semaglutide start) by using the following parameter: HbA1c in mmol/mol
Metabolic health at 6 months after surgery (glucose) | 6 months
  To study metabolic health 6 months after surgery (3 after semaglutide start) by using the following parameter: glucose mmol/l
Metabolic health at 6 months after surgery (triglyceride) | 6 months
  To study metabolic health 6 months after surgery (3 after semaglutide start) by using the following parameter: triglycerides in mmol/l
Metabolic health at 6 months after surgery (LDL) | 6 months
  To study metabolic health 6 months after surgery (3 after semaglutide start) by using the following parameter: LDL in mmol/l
Metabolic health at 6 months after surgery (HDL) | 6 months
  To study metabolic health 6 months after surgery (3 after semaglutide start) by using the following parameter: HDL in mmol/l
Metabolic health at 6 months after surgery (total cholesterol) | 6 months
  To study metabolic health 6 months after surgery (3 after semaglutide start) by using the following parameter: total cholesterol in mmol/l
Metabolic health at 12 months after surgery (bloodpressure) | 12 months
  To study metabolic health 12 months after surgery (9 months after semaglutide start) by using the following parameter: bloodpressure in mmHg
Metabolic health at 12 months after surgery (HbA1c) | 12 months
  To study metabolic health 12 months after surgery (9 months after semaglutide start) by using the following parameter: HbA1c in mmol/mol
Metabolic health at 12 months after surgery (glucose) | 12 months
  To study metabolic health 12 months after surgery (9 months after semaglutide start) by using the following parameter: glucose in mmol/l
Metabolic health at 12 months after surgery (triglyceride) | 12 months
  To study metabolic health 12 months after surgery (9 months after semaglutide start) by using the following parameter: triglycerides in mmol/l
Metabolic health at 12 months after surgery (LDL) | 12 months
  To study metabolic health 12 months after surgery (9 months after semaglutide start) by using the following parameter: LDL in mmol/l
Metabolic health at 12 months after surgery (HDL) | 12 months
  To study metabolic health 12 months after surgery (9 months after semaglutide start) by using the following parameter: HDL in mmol/l
Metabolic health at 12 months after surgery (total cholesterol) | 12 months
  To study metabolic health 12 months after surgery (9 months after semaglutide start) by using the following parameter: total cholesterol in mmol/l
Metabolic health at 18 months after surgery (bloodpressure) | 18 months
  To study metabolic health 18 months after surgery (15 months after semaglutide start) by using the following parameter: bloodpressure in mmHg
Metabolic health at 18 months after surgery (HbA1c) | 18 months
  To study metabolic health 18 months after surgery (15 months after semaglutide start) by using the following parameter: HbA1c in mmol/mol
Metabolic health at 18 months after surgery (glucose) | 18 months
  To study metabolic health 18 months after surgery (15 months after semaglutide start) by using the following parameter: glucose mmol/l
Metabolic health at 18 months after surgery (triglyceride) | 18 months
  To study metabolic health 18 months after surgery (15 months after semaglutide start) by using the following parameter: triglycerides in mmol/l
Metabolic health at 18 months after surgery (LDL) | 18 months
  To study metabolic health 18 months after surgery (15 months after semaglutide start) by using the following parameter: LDL in mmol/l
Metabolic health at 18 months after surgery (HDL) | 18 months
  To study metabolic health 18 months after surgery (15 months after semaglutide start) by using the following parameter: HDL in mmol/l
Metabolic health at 18 months after surgery (total cholesterol) | 18 months
  To study metabolic health 18 months after surgery (15 months after semaglutide start) by using the following parameter: total cholesterol mmol/l
Health-related quality of life also related to gastro intestinal symptoms before surgery | Screening for surgery
  To study health-related quality of life (HRQOL) also related to gastro-intestinal symptoms before surgery (before semaglutide start) using the BODY-Q questionnaire
Health-related quality of life also related to gastro intestinal symptoms 3 months after surgery | 3 months
  To study health-related quality of life (HRQOL) also related to gastro-intestinal symptoms at start of treatment (at semaglutide start) questionnaire
Health-related quality of life also related to gastro intestinal symptoms 6 months after surgery | 6 months
  To study health-related quality of life (HRQOL) also related to gastro-intestinal symptoms 6 months after surgery (3 months after semaglutide start) questionnaire
Health-related quality of life also related to gastro intestinal symptoms | 12 months
  To study health-related quality of life (HRQOL) also related to gastro-intestinal symptoms 12 months after surgery (9 months after semaglutide start) questionnaire
Health-related quality of life also related to gastro intestinal symptoms | 18 months
  To study health-related quality of life (HRQOL) also related to gastro-intestinal symptoms 18 months after surgery (15 months after semaglutide start) questionnaire
Cardiorespiratory fitness level before surgery | Screening for surgery
  To evaluate the change in cardiorespiratory fitness level of the participants before surgery (before semaglutide start ) using a VO2 max test
Cardiorespiratory fitness level 3 months after surgery | 3 months
  To evaluate the change in cardiorespiratory fitness level of the participants 3 months after surgery (at semaglutide start) using a VO2 max test
Cardiorespiratory fitness level 6 months after surgery | 6 months
  To evaluate the change in cardiorespiratory fitness level of the participants 6 months after surgery (3 months after semaglutide start) using a VO2 max test
Cardiorespiratory fitness level 12 months after surgery | 12 months
  To evaluate the change in cardiorespiratory fitness level of the participants 12 months after surgery (9 months after semaglutide start) using a VO2 max test
Cardiorespiratory fitness level 18 months after surgery | 18 months
  To evaluate the change in cardiorespiratory fitness level of the participants 18 months after surgery (15 months after semaglutide start) using a VO2 max test
Change in liver fat and liver stiffness at start of treatment | Screening for study
  To study the change in liver fat and liver stiffness, measured with vibration controlled transient elastography, at start of treatment with semaglutide
Change in liver fat and liver stiffness 15 months after semaglutide start | 15 months
  To study the change in liver fat and liver stiffness, measured with vibration controlled transient elastography, 15 months after semaglutide start
To describe the persistence of therapy | 15 months
  The number of patients who persisted the therapy given in the study
To describe the average weekly dose | 15 months
  The number of patient on all possible dosages at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Greve, prof, Principal Investigator — Zuyderland Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646
- [Background] Bray GA, Fruhbeck G, Ryan DH, Wilding JP. Management of obesity. Lancet. 2016 May 7;387(10031):1947-56. doi: 10.1016/S0140-6736(16)00271-3. Epub 2016 Feb 10. PMID 26868660
- [Background] Busetto L, Dicker D, Azran C, Batterham RL, Farpour-Lambert N, Fried M, Hjelmesaeth J, Kinzl J, Leitner DR, Makaronidis JM, Schindler K, Toplak H, Yumuk V. Practical Recommendations of the Obesity Management Task Force of the European Association for the Study of Obesity for the Post-Bariatric Surgery Medical Management. Obes Facts. 2017;10(6):597-632. doi: 10.1159/000481825. Epub 2017 Dec 6. PMID 29207379
- [Background] Apovian CM, Aronne LJ, Bessesen DH, McDonnell ME, Murad MH, Pagotto U, Ryan DH, Still CD; Endocrine Society. Pharmacological management of obesity: an endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2015 Feb;100(2):342-62. doi: 10.1210/jc.2014-3415. Epub 2015 Jan 15. PMID 25590212
- [Background] Nuffer W, Trujillo JM, Megyeri J. A Comparison of New Pharmacological Agents for the Treatment of Obesity. Ann Pharmacother. 2016 May;50(5):376-88. doi: 10.1177/1060028016634351. Epub 2016 Feb 17. PMID 26887340
- [Background] Madsbad S, Dirksen C, Holst JJ. Mechanisms of changes in glucose metabolism and bodyweight after bariatric surgery. Lancet Diabetes Endocrinol. 2014 Feb;2(2):152-64. doi: 10.1016/S2213-8587(13)70218-3. Epub 2014 Feb 3. PMID 24622719
- [Background] Sjostrom L. Review of the key results from the Swedish Obese Subjects (SOS) trial - a prospective controlled intervention study of bariatric surgery. J Intern Med. 2013 Mar;273(3):219-34. doi: 10.1111/joim.12012. Epub 2013 Feb 8. PMID 23163728
- [Background] Gloy VL, Briel M, Bhatt DL, Kashyap SR, Schauer PR, Mingrone G, Bucher HC, Nordmann AJ. Bariatric surgery versus non-surgical treatment for obesity: a systematic review and meta-analysis of randomised controlled trials. BMJ. 2013 Oct 22;347:f5934. doi: 10.1136/bmj.f5934. PMID 24149519
- [Background] Reges O, Greenland P, Dicker D, Leibowitz M, Hoshen M, Gofer I, Rasmussen-Torvik LJ, Balicer RD. Association of Bariatric Surgery Using Laparoscopic Banding, Roux-en-Y Gastric Bypass, or Laparoscopic Sleeve Gastrectomy vs Usual Care Obesity Management With All-Cause Mortality. JAMA. 2018 Jan 16;319(3):279-290. doi: 10.1001/jama.2017.20513. PMID 29340677
- [Background] Sjostrom L, Peltonen M, Jacobson P, Sjostrom CD, Karason K, Wedel H, Ahlin S, Anveden A, Bengtsson C, Bergmark G, Bouchard C, Carlsson B, Dahlgren S, Karlsson J, Lindroos AK, Lonroth H, Narbro K, Naslund I, Olbers T, Svensson PA, Carlsson LM. Bariatric surgery and long-term cardiovascular events. JAMA. 2012 Jan 4;307(1):56-65. doi: 10.1001/jama.2011.1914. PMID 22215166
- [Background] Colquitt JL, Picot J, Loveman E, Clegg AJ. Surgery for obesity. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003641. doi: 10.1002/14651858.CD003641.pub3. PMID 19370590
- [Background] Karmali S, Brar B, Shi X, Sharma AM, de Gara C, Birch DW. Weight recidivism post-bariatric surgery: a systematic review. Obes Surg. 2013 Nov;23(11):1922-33. doi: 10.1007/s11695-013-1070-4. PMID 23996349
- [Background] Tettero OM, Monpellier VM, Janssen IMC, Steenhuis IHM, van Stralen MM. Early Postoperative Weight Loss Predicts Weight Loss up to 5 Years After Roux-En-Y Gastric Bypass, Banded Roux-En-Y Gastric Bypass, and Sleeve Gastrectomy. Obes Surg. 2022 Sep;32(9):2891-2902. doi: 10.1007/s11695-022-06166-x. Epub 2022 Jul 16. PMID 35842505
- [Background] Mor A, Sharp L, Portenier D, Sudan R, Torquati A. Weight loss at first postoperative visit predicts long-term outcome of Roux-en-Y gastric bypass using Duke weight loss surgery chart. Surg Obes Relat Dis. 2012 Sep-Oct;8(5):556-60. doi: 10.1016/j.soard.2012.06.014. Epub 2012 Jul 16. PMID 22920966
- [Background] Pinto-Bastos A, Conceicao EM, Machado PPP. Reoperative Bariatric Surgery: a Systematic Review of the Reasons for Surgery, Medical and Weight Loss Outcomes, Relevant Behavioral Factors. Obes Surg. 2017 Oct;27(10):2707-2715. doi: 10.1007/s11695-017-2855-7. PMID 28791623
- [Background] RJ Rosenthal. Failure of weight loss or weight regain after bariatric surgery. Bariatric Times. 2012.
- [Background] McKenna D, Selzer D, Burchett M, Choi J, Mattar SG. Revisional bariatric surgery is more effective for improving obesity-related co-morbidities than it is for reinducing major weight loss. Surg Obes Relat Dis. 2014 Jul-Aug;10(4):654-9. doi: 10.1016/j.soard.2013.12.007. Epub 2013 Dec 18. PMID 24708909
- [Background] Brethauer SA, Kothari S, Sudan R, Williams B, English WJ, Brengman M, Kurian M, Hutter M, Stegemann L, Kallies K, Nguyen NT, Ponce J, Morton JM. Systematic review on reoperative bariatric surgery: American Society for Metabolic and Bariatric Surgery Revision Task Force. Surg Obes Relat Dis. 2014 Sep-Oct;10(5):952-72. doi: 10.1016/j.soard.2014.02.014. Epub 2014 Feb 22. PMID 24776071
- [Background] Christou GA, Katsiki N, Blundell J, Fruhbeck G, Kiortsis DN. Semaglutide as a promising antiobesity drug. Obes Rev. 2019 Jun;20(6):805-815. doi: 10.1111/obr.12839. Epub 2019 Feb 15. PMID 30768766
- [Background] Shaefer CF Jr, Kushner P, Aguilar R. User's guide to mechanism of action and clinical use of GLP-1 receptor agonists. Postgrad Med. 2015;127(8):818-26. doi: 10.1080/00325481.2015.1090295. Epub 2015 Sep 15. PMID 26371721
- [Background] Wadden TA, Bailey TS, Billings LK, Davies M, Frias JP, Koroleva A, Lingvay I, O'Neil PM, Rubino DM, Skovgaard D, Wallenstein SOR, Garvey WT; STEP 3 Investigators. Effect of Subcutaneous Semaglutide vs Placebo as an Adjunct to Intensive Behavioral Therapy on Body Weight in Adults With Overweight or Obesity: The STEP 3 Randomized Clinical Trial. JAMA. 2021 Apr 13;325(14):1403-1413. doi: 10.1001/jama.2021.1831. PMID 33625476
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Background] Rubino D, Abrahamsson N, Davies M, Hesse D, Greenway FL, Jensen C, Lingvay I, Mosenzon O, Rosenstock J, Rubio MA, Rudofsky G, Tadayon S, Wadden TA, Dicker D; STEP 4 Investigators. Effect of Continued Weekly Subcutaneous Semaglutide vs Placebo on Weight Loss Maintenance in Adults With Overweight or Obesity: The STEP 4 Randomized Clinical Trial. JAMA. 2021 Apr 13;325(14):1414-1425. doi: 10.1001/jama.2021.3224. PMID 33755728